CLINICAL TRIAL: NCT05835349
Title: A Real-World Evidence Observational Study of VenusP-ValveTM System in the Treatment of Patients with Native RVOT Dysfunction
Brief Title: Observational Study of Venus P-Valve
Acronym: Registry
Status: Recruiting | Type: Observational
Sponsor: Venus MedTech (HangZhou) Inc. (Industry)
Collaborators: IQVIA MedTech BV of Antwerp, Belgium (Unknown); MDCECRO LLC (Network)
Responsible Party: Sponsor
Other Study IDs: VTPR-22-08
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Right Ventricular Outflow Tract Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: transcatheter pulmonary valve implantation (TPVI) — A stent-mounted valve is introduced over a guidewire and positioned in the RVOT, followed by balloon inflation to deploy the valve.

SUMMARY:
Real-world evidence, retrospective and prospective, non-randomized, multicenter observational study of VenusP-ValveTM System in treating moderate or greater pulmonary regurgitation with/without pulmonary stenosis in patients with native right ventricular outflow tract (RVOT).

DETAILED DESCRIPTION:
All subjects will be followed up through five years for the observed outcome measures, which will be analyzed and reported to regulatory authorities as required.

Post-procedure, a clinical visit will be scheduled at discharge, thirty days, six months, one year, and annually thereafter to five years.

ELIGIBILITY:
Inclusion Criteria

1. Patients with native RVOT (including transvalvular patch repair) are present with moderate or greater pulmonary regurgitation with/without stenosis and are clinically indicated for pulmonary valve intervention.
2. The patient (or the patient's legally authorized representative) is willing to consent to participate in the study and will commit to completing all follow-up requirements.

Exclusion Criteria:

1. Patients with any condition contraindicated by the IFU or inability to comply with the Venus P-ValveTM System Instructions for Use or the study protocol.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Baseline enrolment criteria
  * 12 years old up to 70 years old
  * Weight ≥ 30kg
  * With evidence of moderate or severe (≥3+) pulmonary regurgitation by Transthoracic Echocardiography (TTE)
  * With >30% pulmonary regurgitation fraction as defined by cardiac Magnetic Resonance Imaging (MRI)
  * The subject is symptomatic from his/her pulmonary regurgitation or meets MRI criteria for intervention Right Ventricular Ejection Fraction (RVEF) < 45%, Pulmonary Regurgitant Fraction (PRRF) >30% and increased Right Ventricular End Diastolic Volume (RVEDV) Index (RVEDVI) >150mL/m²
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Non-hierarchical composite endpoint | at six months
  * Freedom from VenusP-ValveTM (catheter or surgical) reintervention
  * Acceptable hemodynamic function, defined as:
    1. Mild or less regurgitation measured by echocardiography; AND
    2. Mean RVOT gradient as measured by echocardiography ≤35mmHg.

SECONDARY OUTCOMES:
Procedural Success | at 30 days
  Procedure success at 30 days, defined as:
  * Freedom from procedure/device-related mortality
  * Freedom from Venus P-ValveTM (catheter or surgical) reintervention concerning index procedure or device
  * Acceptable hemodynamic function
  * Original intended valve in situ
Occurrence of Events | through five years
  Occurrence of the following events through 5 years of follow-up:
  * All-cause mortality and procedure/device-related mortality
  * Venus P-ValveTM (catheter or surgical) reintervention
  * Venus P-ValveTM dysfunction
  * Serious procedure/device-related adverse events
Functional status | through five years
  New York Heart Association (NYHA) classification out to 5 years
Health-state utility score | through five years
  Health-state utility score as measured by the EQ-5D at pre-implant, 30 days, 6 months, 1 year and annually thereafter through 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Shakeel A. Qureshi, MD, Principal Investigator — Evelina Children's Hospital
Locations (10):
- France (4):
  - CHU Bordeaux, Pessac, Nouvelle-Aquitaine
  - Chu Nantes, Nantes, Pays de la Loire Region
  - Marie Lannelongue, Le Plessis-Robinson, Île-de-France Region
  - Hopital Necker-Enfants malades, Paris, Île-de-France Region
- Germany (2):
  - Heart CenterMunich, Munich, Bavaria
  - Clinic of Congenital Heart Disease, Berlin, State of Berlin
- Italy (2):
  - OPBG Rome, Rome, Lazio
  - S. Donato Milan, Milan, Lombardy
- United Kingdom (2):
  - Leeds General Infirmary, Leeds, England
  - Evelina Children's Hospital, London, England

IPD SHARING:
Plan to Share IPD: No
Under attention to laws and regulations concerning personal data protection, empirical (non personally identifiable) data is anticipated to be shared within the clinical investigator team. Processed and analysed data would be shared within a wider community of medical professionals through professional conference presentations and peer-reviewed journal publications.